CLINICAL TRIAL: NCT00641654
Title: An Open-label Multicenter Study Evaluating the Efficacy and Safety of 24 or 48 Weeks Pegylated Interferon Alfa-2a 40 kD (PEGASYS) Combination Therapy With Ribavirin (Copegus) in Patients With Chronic Hepatitis C Genotype 2 or 3 Infection Who Previously Have Relapsed After a Minimum of 12 Weeks and a Maximum of 24 Weeks of Therapy With Pegylated Interferon and Ribavirin
Brief Title: Combination Therapy With Pegylated Interferon and Ribavirin in Patients With Chronic Hepatitis C Genotype 2 or 3 Infection Who Previously Have Relapsed After Therapy With Pegylated Interferon and Ribavirin
Acronym: RelapC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment problems in Denmark and Norway
Sponsor: Göteborg University (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudractCT 2006-003409-18
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; genotype 2 or 3; relapse; pegylated interferon; ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic; Recurrence | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Patients having previously received 24 weeks of therapy with pegylated interferon and ribavirin will be treated with pegylated interferon alfa-2a kD (PEGASYS) plus ribavirin, (Copegus) for a treatment period of 48 weeks, with a follow-up period of 24 weeks irrespective of the level of HCV-RNA measured in plasma on treatment day 27.
  Interventions: Drug: Pegylated interferon alfa-2a and ribavirin
- B (Active Comparator): Patients having previously received less than 24 weeks but at least 12 weeks of therapy with pegylated interferon and Ribavirin and having detectable HCV-RNA in a plasma sample obtained on treatment day 27 (i.e. the day before the 5th dose of pegylated interferon in this study) as analyzed by means of COBAS TaqMan 48TM will be treated with pegylated interferon alfa-2a KD (PEGASYS®) plus ribavirin, (Copegus®) for a treatment period of 48 weeks, with a follow-up period of 24 weeks.
  Interventions: Drug: Pegylated interferon alfa-2a and ribavirin
- C (Active Comparator): Patients having previously received less than 24 weeks but at least 12 weeks of therapy with pegylated interferon and Ribavirin and having undetectable HCV-RNA in a plasma sample obtained on treatment day 27 (i.e. the day before the 5th dose of pegylated interferon in this study) as analyzed by means of COBAS TaqMan 48TM will be treated with pegylated interferon alfa-2a KD (PEGASYS®) plus ribavirin, (Copegus®) for a treatment period of 24 weeks, with a follow-up period of 24 weeks.
  Interventions: Drug: Pegylated interferon alfa-2a and ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a and ribavirin — Arm A: Pegylated interferon alfa-2a Injection, 180 µg sc x 1/w for 48 weeks Ribavirin Tablet 200 mg weight based 5 or 6 per day for 48 weeks
  Other Names: Pegasys; Copegus
  Arms: A
Drug: Pegylated interferon alfa-2a and ribavirin — Arm B:Pegylated interferon alfa-2a Injection, 180 µg sc x 1/w for 48 weeks Ribavirin Tablet 200 mg weight based 5 or 6 per day for 48 weeks
  Other Names: Pegasys; Copegus
  Arms: B
Drug: Pegylated interferon alfa-2a and ribavirin — Arm C:Pegylated interferon alfa-2a Injection, 180 µg sc x 1/w for 24 weeks Ribavirin Tablet 200 mg weight based 5 or 6 per day for 24 weeks
  Other Names: Pegasys; Copegus
  Arms: C

SUMMARY:
To evaluate the efficacy of pegylated interferon alfa-2a 40 kD (PEGASYS) combination therapy with ribavirin (Copegus)given for 24 or 48 weeks in patients with chronic hepatitis C (CHC) virus infection genotype 2 or 3 who responded during (i.e. had HCV-RNA <50 IU/mL at the end of previous therapy), but relapsed after (i.e. had detectable HCV-RNA after the end of prior treatment) previous therapy with pegylated interferon and ribavirin given for at least 12 weeks and at most 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Serum HCV-RNA ≥ 15 IU/mL. HCV genotype 2 or/and 3 infection confirmed within the past 6 months preceding the initiation of test drug dosing. The HCV genotype must have been reconfirmed after the termination of the previous treatment period
* Previous relapse (i.e. HCV-RNA < 50 IU/mL at end of previous therapy) after one treatment period with pegylated interferon alfa-2a or alfa-2b combination therapy with ribavirin for at least 12 weeks and at most 24 weeks
* A minimum of 24 weeks must have elapsed since the last dose of pegylated interferon or ribavirin in the previous treatment period before the patients can be included in this study
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Patients with suspected cirrhosis or transition to cirrhosis must have an abdominal ultrasound, CT scan, or MRI scan without evidence of hepatocellular carcinoma and a serum AFP < 100 ng/mL within 2 months of randomization
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using effective contraception during treatment and during the 6 months after treatment end
* Having a liver biopsy obtained within 5 years of this study is encouraged, but optional in accordance with local treatment traditions.

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Previous non-response during treatment (as defined as having detectable HCV RNA ≥ 50 IU/ml at the end of previous treatment) with pegylated interferon alfa-2a or alfa-2b combination therapy with ribavirin for at least 12 weeks and at most 24 weeks
* Less than 24 weeks have elapsed since the last dose of pegylated interferon or ribavirin in the previous treatment period prior to inclusion in this study.
* Therapy with any systemic anti-viral

  * anti-neoplastic
  * immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤ 6 months prior to the first dose of study drug
* Any investigational drug ≤ 6 weeks prior to the first dose of study drug. HCV genotype 1, 4, 5 or 6 infection
* Positive test at screening for anti-HAV IgM Ab

  * HBsAg
  * anti-HBc IgM Ab
  * anti-HIV Ab
* Evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History or other evidence of decompensated liver disease
* Neutrophil count < 1500 cells/mm3 or platelet count < 75,000 cells/mm3 at screening
* Serum creatinine level > 2 mg/dl (> 124 µmol/L) or creatinine clearance < 50 ml/minute at screening
* Severe psychiatric disease, especially depression, as judged by the treating physician
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease

  * severe chronic pulmonary disease associated with functional limitation
  * severe cardiac disease
  * major organ transplantation or other evidence of severe illness
  * malignancy
  * any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Thyroid dysfunction not adequately controlled (TSH and T4 levels out of normal range)
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration) or

  * clinically relevant ophthalmological disorder due to diabetes mellitus or
  * hypertension
* Evidence of drug abuse (including excessive alcohol consumption) in accordance with local therapeutic traditions. (Patients receiving Methadone or Subutex therapy may be included in this study.)
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Hemoglobin < 11.3 g/dL (< 7.0 mmol/L) in women or < 12.9 g/dL (< 8.0 mmol/L) in men at screening.
* Any patient with an increased baseline risk for anemia (e.g. thalassemia, spherocytosis, etc) or for whom anemia would be medically problematic
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sustained viral response (SVR) rate defined as percentage of patients with non-detectable HCV-RNA 24 weeks after completion of the 24 or 48 week treatment period. | 24 weeks after completion of the 24 or 48 week treatment period.

SECONDARY OUTCOMES:
Sustained viral response (SVR)rate and percentage of patients with normal serum ALT levels and its association with prespecified factors e.g. viral load | 24 weeks after complection of the 24 or 48 week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar PE Norkrans, MD Prof, Principal Investigator — Sahlgrenska University Hospital,Göteborg University
Locations (1):
- Dept of Infectious Diseases, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Lagging M, Rembeck K, Rauning Buhl M, Christensen P, Dalgard O, Farkkila M, Hellstrand K, Langeland N, Lindh M, Westin J, Norkrans G. Retreatment with peg-interferon and ribavirin in patients with chronic hepatitis C virus genotype 2 or 3 infection with prior relapse. Scand J Gastroenterol. 2013 Jul;48(7):839-47. doi: 10.3109/00365521.2013.793389. PMID 23795661